CLINICAL TRIAL: NCT01645852
Title: A Randomized Phase II Study of the Effect of a Low Calorie Diet on Patients Undergoing Liver Resection
Brief Title: A Phase II Study of the Effect of a Low Calorie Diet on Patients Undergoing Liver Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DMS 12052
Record Dates: First submitted 2012-07-17; First posted 2012-07-20 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Nonalcoholic Fatty Liver Disease; Hepatic Steatosis; Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): No specified diet for one week prior to hepatic resection.
- Low calorie diet (Active Comparator): Low calorie diet (five units of Optifast 800 {Nestle Nutrition, Vevey, Switzerland} plus an unlimited volume of calorie free fluids per day) for one week prior to hepatic resection.
  Interventions: Dietary Supplement: Optifast 800

INTERVENTIONS:
Dietary Supplement: Optifast 800 — Five units of Optifast 800 plus an unlimited volume of calorie-free fluids per day for one week prior to hepatic resection.
  Arms: Low calorie diet

SUMMARY:
The purpose of this study is to measure the effect of a short-term low calorie diet on patients with a Body Mass Index (BMI) over 25 who are undergoing liver surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Clinical indication for a therapeutic liver resection
* BMI of 25 kg/m2 or greater
* Informed Consent

Exclusion Criteria:

* Inability to comply with the pre-op diet
* Patients who have lost 5% or more of their usual body weight over the preceding one month
* Female patients of childbearing age who have a positive pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The effect of a low calorie diet on intra-operative blood loss, technical ease of hepatic transection, complication rates (including infectious complications), length of stay and mortality in patients undergoing liver surgery. | 30 days post-operatively
  Intra-operative blood loss will be strictly quantified. Units of autologous or donor blood transfused will be recorded. The surgeon will assess the ease of liver mobilization and parenchymal transection using a 1-5 scale where 1 is easy and 5 is hard. Post-operative complications, length of stay and mortality will be recorded.

SECONDARY OUTCOMES:
The effect of a low calorie diet on steatosis and steatohepatitis. | 30 days post-operatively
  Using tissue from hepatic parenchyma adjacent to resected neoplasms steatosis and steatohepatitis will be evaluated by a pathologist blinded to dietary intervention. Steatosis will be defined as mild, moderate or severe if 5-33%, 34-66%, or >66% of hepatocytes contain fat inclusions. Steatohepatitis will be defined using NAFLD (Non-Alcoholic Fatty Liver Disease) Activity Score (NAS) as an NAS 4 or greater, with <4 defined as no steatohepatitis.
The mechanism of decreased steatosis in patients undergoing a low-calorie pre-op diet by measuring levels of expression of molecules involved in the de novo synthesis, hepatic uptake and degradation of lipids. | 30 days post-operatively
  Levels of expression of molecules involved in the de novo synthesis, hepatic uptake and degradation of lipids will be measured to evaluate the mechanism of decreased steatosis.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Barth, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (3):
- United States (3):
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Fletcher Allen Health Care, Burlington, Vermont